CLINICAL TRIAL: NCT00680862
Title: Qualitative Assessment of Implementing Routine Rapid HIV Testing
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: SHP 08-158
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infections
Keywords: HIV; screening
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1: VA employees

SUMMARY:
Qualitative assessment of implementing routine HIV rapid testing in primary care clinics within VA

DETAILED DESCRIPTION:
Background:

During the past three decades, human immunodeficiency virus (HIV) infection and acquired immunodeficiency syndrome (AIDS) have caused extensive illness and death in the United States. Since the advent of the HIV epidemic, the VA healthcare system has been significantly impacted. Veterans are at much higher HIV risk than the general population. In addition, a significant proportion of VA patients are members of minority groups, and are homeless, both patient categories which have also been linked to high HIV prevalence. Because the VA is the largest provider of HIV treatment in the US, it is imperative that researchers develop innovative methods to 1) identify HIV-positive individuals, 2) provide them with the knowledge of their HIV-positive status; 3) do so early enough in the disease so that patients can be placed into care, so that antiretroviral therapies can be effective, and the HIV epidemic can be slowed and reversed.

Current HIV testing methods have been highly ineffective in this regard, due in large measure to the method itself. Conventional HIV testing requires both a blood draw and laboratory analysis, requiring a patient to schedule a future visit to receive results. Consequently, a significant number of people simply do not return for their test results. Current HIV prevalence figures bear this out. The Centers for Disease Control and Prevention (CDC) estimates that of the 1.2 million HIV infected persons in the US, as many as 1/3 are unaware of their infection. Indeed, the CDC now recommends routine HIV testing for all Americans. This recommendation was predicated on the evidence that moving from a risk-based, to a routine testing model is one of the most effective ways to significantly increase testing rates. As better HIV identification systems begin to spread through the VHA, the VHA must determine the proper place for broader routine HIV rapid testing programs in their delivery systems. Demonstrating effectiveness is only the first step. To make policy recommendations, we must better understand the challenges of implementing a testing system that would apply to all, not just at-risk patients.

The move toward routine HIV testing, combined with a novel diagnostic tool (rapid testing) although highly effective, provides many implementation challenges. For example, what are the unintended adverse consequences in implementing NRT? What are the barriers and facilitators to implementation? How important are local nursing and physician champions and opinion leaders? These issues are of paramount importance in reaching an evidence-based consensus as to what a 'best practices' approach could look like within a large, decentralized healthcare organization like VA.

Objectives:

The specific aims of this project then, are:

1. To develop generalized qualitative methods and instruments which can be used to evaluate VA HIV rapid testing implementation efforts;
2. To employ these developed instruments to qualitatively document the implementation of our previously successful NRT strategy for spreading NRT to VA primary/urgent care practice at our downtown Los Angeles Outpatient Clinic (OPC);
3. To explore and document barriers, facilitators, and unintended consequences of implementing our NRT model of HIV testing at LAOPC.

Methods:

We used qualitative methods to conduct formative and process evaluations which allowed us to fully assess our research objective, which were:

A thorough examination, exploration and description of the barriers and facilitators to implementing NRT at the Los Angeles Outpatient Clinic (OPC).

Status:

project objectives completed; manuscript being developed

ELIGIBILITY:
Inclusion Criteria:

- VA employees of LA OPC who are involved in HIV care and/or policy

Exclusion Criteria:

- n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: key informant VA employees
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Anaya, PhD MA, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

REFERENCES:
- [Result] Anaya HD, Bokhour B, Feld J, Golden JF, Asch SM, Knapp H. Implementation of routine rapid HIV testing within the U.S. Department of Veterans Affairs Healthcare System. J Healthc Qual. 2012 Sep-Oct;34(5):7-14. doi: 10.1111/j.1945-1474.2011.00151.x. Epub 2011 May 25. PMID 22060061

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: VA employees
Arm/Group | Group 1
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed the Survey
Description: survey responses from participants on thoughts pertaining to implementation of HIV rapid testing
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 25
participants | 25

ADVERSE EVENTS:
Description: Serious and other [non-serious] adverse events were not collected or assessed as part of the study
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes